CLINICAL TRIAL: NCT05348577
Title: A Phase III Double-Blind, Randomised, Placebo-Controlled Study Assessing the Efficacy and Safety of Capivasertib + Docetaxel Versus Placebo + Docetaxel as Treatment for Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: Study of Capivasertib + Docetaxel vs Placebo + Docetaxel as Treatment for Metastatic Castration Resistant Prostate Cancer (mCRPC)
Acronym: CAPItello280
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D361EC00001; 2023-504996-26-00 (Registry Identifier: CTIS); 2021-005201-27 (EudraCT Number)
Record Dates: First submitted 2022-03-18; First posted 2022-04-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer,; metastatic; castration resistant; capivasertib,; AKT inhibitor,; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — capivasertib; Docetaxel

STUDY DESIGN:
Intervention Model Description: Approximately 1350 participants will be enrolled and screened to achieve a total of approximately 1000 assigned in a 1:1 ratio to one of the two parallel groups to receive either capivasertib or placebo, in combination with docetaxel on a background of ADT for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blinded, neither the patients nor the investigator will know what study intervention was assigned.
  Capivasertib and placebo film-coated tablets will be identical in appearance and presented in the same packaging to ensure blinding of the capivasertib.
  All personnel involved with the statistical analysis of the study will remain blinded until database lock and CSP deviations have been identified.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- capivasertib + docetaxel (Experimental): Participants receive capivasertib in combination with docetaxel and steroids on a background of ADT.
  Interventions: Drug: capivasertib; Drug: docetaxel
- placebo + docetaxel (Placebo Comparator): Participants receive placebo in combination with docetaxel and steroids on a background of ADT.
  Interventions: Drug: docetaxel; Other: placebo

INTERVENTIONS:
Drug: capivasertib — 320 mg (2 tablets) BD given on an intermittent weekly dosing schedule. Patients will be dosed on Days 2 to 5, 9 to 12, and 16 to 19 in each week of a 21-day treatment cycle.
  Number of Cycles: until disease progression or unacceptable toxicity develops, death, or if the patient requests to stop the study treatment.
  Arms: capivasertib + docetaxel
Drug: docetaxel — Patients will receive docetaxel in intravenous infusion, 75 mg/m2 BSA, on Day 1 of the 21-day cycles for up to 6 to 10 cycles, according to standard of care practices.
Other: placebo — matched to capivasertib appearance (2 tablets) BD given orally on an intermittent weekly dosing schedule. Patients will be dosed on Days 2 to 5, 9 to 12, and 16 to 19 in each week of a 21-day treatment cycle. Number of Cycles: until disease progression or unacceptable toxicity develops, death, or if the patient requests to stop the study treatment.
  Arms: placebo + docetaxel

SUMMARY:
This study will assess the efficacy and safety of capivasertib plus docetaxel versus placebo plus docetaxel in participants with metastatic castration resistant prostate cancer (mCRPC), all participants will receive the docetaxel with steroid therapy and receive androgen deprivation therapy. The intention of the study is to demonstrate that the combination of capivasertib plus docetaxel is superior to placebo plus docetaxel with respect to the overall survival and/or the radiographic progression free survival of study participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed prostate adenocarcinoma without predominant neuroendocrine or small cell cancers
* Metastatic disease documented prior to randomisation by clear evidence of ≥ 1 bone lesion (defined as 1 lesion with positive uptake on bone scan) and/or ≥ 1 soft tissue lesion (measurable or non-measurable)
* Patient must have been previously treated with a next generation hormonal agent (NHA), ie, abiraterone, enzalutamide, apalutamide or darolutamide, for prostate cancer for at least 3 months and shown evidence of disease progression (radiological or via PSA assessment) while receiving the NHA
* Evidence of mCRPC with progression of disease despite androgen deprivation therapy (ADT)
* Serum testosterone level ≤ 50 ng/dL
* Candidate for docetaxel and steroid therapy
* Ongoing ADT with LHRH agonist, LHRH antagonist, or bilateral orchiectomy
* Eastern Cooperative Oncology Group (ECOG)/World Health Organisation (WHO) performance status 0 to 1 and anticipated minimum life expectancy of 12 weeks
* Confirmation that archival formalin-fixed paraffin-embedded (FFPE) tumour tissue sample which meets the minimum pathology and sample requirements is available to send to the central laboratory
* Able and willing to swallow and retain oral medication
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Radiotherapy with a wide field of radiation within 4 weeks before start of study treatment
* Major surgery (excl. placement of vascular access, transurethral resection of prostate, bilateral orchiectomy, internal stents) within 4 weeks of start of study treatment
* Brain metastases,or spinal cord compression (unless spinal cord compression is asymptomatic and stable and not requiring steroids for at least 4 weeks prior to start of study treatment)
* Any of the following cardiac criteria:

  i. Mean resting corrected QT interval (QTc) >470 msec from 3 consecutive ECGs ii. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG iii. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age,or any concomitant medication known to prolong the QT interval iv. Experience of any of the following procedures or conditions in the preceding 3 months: coronary artery bypass graft, vascular stent, myocardial infarction, unstable angina pectoris, congestive heart failure NYHA Grade ≥2 v. Symptomatic hypotension - systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg vi. haemodinamic instability
* Clinically significant abnormalities of glucose metabolism as defined by any of the following:

  i. Patients with diabetes mellitus (DM) type 1 or DM type 2 requiring insulin treatment ii. HbA1c ≥8.0% (63.9 mmol/mol)
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  i. Absolute neutrophil count < 1.5x 10^9/L ii. Platelet count < 100x 10^9/L iii. Haemoglobin < 9 g/dL (< 5.59 mmol/L) iv. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5x upper limit of normal (ULN) if no demonstrable liver metastases or > 5x ULN in the presence of liver metastases. Elevated alkaline phosphatase (ALP) is not exclusionary if due to the presence of bone metastases and liver function is otherwise considered adequate in the investigator's judgement v. Total bilirubin > 1.5x ULN (participants with confirmed Gilbert's syndrome may be included in the study with a higher value) vi. Creatinine clearance < 50 mL/min per the Cockcroft and Gault formula without the need for chronic dialysis;
* As judged by the investigator, any evidence of diseases (including severe or uncontrolled systemic diseases, uncontrolled hypertension, history of interstitial pneumonia / pneumonitis or interstitial lung disease, renal transplant and active bleeding diseases), which, in the investigator's opinion, makes it undesirable for the patient to participate in the study or that would jeopardise compliance with the protocol.
* Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection, or other condition that would preclude adequate absorption of capivasertib
* Any other disease, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contra-indicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent. Evidence of dementia, altered mental status, or any psychiatric condition that would prohibit understanding or rendering of informed consent.
* Previous allogeneic bone marrow transplant or solid organ transplant
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include adequately resected non-melanoma skin cancer and curatively treated in situ disease.
* Persistent toxicities (CTCAE Grade ≥2) caused by previous anticancer therapy, excluding alopecia. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention in the opinion of the investigator may be included (eg, hearing loss)
* Known to have active hepatitis infection.
* Known to have human immunodeficiency virus (HIV) with a detectable viral RNA load or a CD4+ T-cell count < 350 cells/uL or a history of an acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months, or receiving anti-HIV medications for less than 4 weeks.
* Known to have active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
* Treatment with any of the following:

  i. Prior chemotherapy for CRPC. Chemotherapy for metastatic or localized HSPC (including docetaxel) is allowed provided that chemotherapy was completed ≥ 6months before randomisation and progression of the prostate cancer occurred ≥ 6months after the completion of therapy.

ii. Prior exposure to AKT inhibitors or PI3K inhibitors iii. Any investigational agents or study drugs from a previous clinical study within 30 days or 5 half-lives (whichever is longer) of the first dose of study treatment iv. Any other immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents (except ADT) within 3 weeks of the first dose of study treatment v. Strong inhibitors or strong inducers of cytochrome P450 (CYP)3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort), vi.Use of any live vaccine administration 30 days prior to the initiation of study treatment, during, and for at least 90 days after the last dose of the study treatment

* Drugs known to significantly prolong the QT interval and associated with Torsade de Pointes within 5 half-lives of the first dose of study treatment
* History of hypersensitivity to active or inactive excipients of capivasertib, docetaxel, or drugs with a similar chemical structure or class
* Any restriction or contraindication based on the local prescribing information that would prohibit the use of docetaxel

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in the overall population | up to approximately 46 months
  Overall survival is defined as time from randomisation until the date of death due to any cause.
Radiographic Progression-free Survival (rPFS) in the overall population | up to approximately 37 months
  Radiographic Progression-free Survival (rPFS) is defined as time from randomization to radiographic progression as assessed by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) for soft tissue and/or Prostate Cancer Working Group 3 (PCWG3) for bone or death due to any cause

SECONDARY OUTCOMES:
Overall Survival (OS) in patients with mCRPC and PTEN-proficient tumours (IHC) | up to approximately 46 months
  OS is defined as time from randomisation until the date of death due to any cause.
Overall Survival (OS) in patients with mCRPC and PTEN-deficient tumours (IHC). | up to approximately 46 months
  OS is defined as time from randomisation until the date of death due to any cause.
Radiographic Progression-free Survival (rPFS) in patients with mCRPC and PTEN-proficient tumours (IHC) | up to approximately 37 months
  Radiographic progression-free survival is defined as the time from randomisation to radiographic progression, as assessed by the investigator at local site per RECIST version 1.1 (soft tissue) and/or PCWG3 criteria (bone), or death due to any cause.
Radiographic Progression-free Survival (rPFS) in patients with mCRPC and PTEN-deficient tumours (IHC) | up to approximately 37 months
  Radiographic progression-free survival is defined as the time from randomisation to radiographic progression, as assessed by the investigator at local site per RECIST version 1.1 (soft tissue) and/or PCWG3 criteria (bone), or death due to any cause.
Time to pain progression (TTPP) in the overall population | up to approximately 37 months
  Time to pain progression (TTPP) based on a 2-point increase from baseline in the Brief Pain Inventory-Short Form (BPI-SF) Item 3 'pain at its worse in the last 24 hours' score (scale from 0 ["no pain"] to 10 ["pain as bad as you can imagine"]) and/or initiation of/increase in opioid analgesic use.
Time to first Symptomatic Skeletal-Related Event (SSRE) in the overall population | up to approximately 46 months
  SSRE is defined as time from randomisation until any of the following: use of radiation therapy to prevent or relieve skeletal symptoms; Occurrence of new symptomatic pathological bone fractures; Occurrence of spinal cord compression; Orthopaedic surgical intervention for bone metastasis
Time to deterioration in urinary symptoms (TTDUS) in the overall population | up to approximately 37 months
  Time to deterioration in urinary symptoms (TTDUS) is defined as time from randomization until the change from baseline reaches a clinically meaningful deterioration threshold using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Prostate Questionnaire Urinary Symptoms (QLQ-PR25 (US)) subscale score (EORTC IL166), where the question responses are provided on a numerical rating scale ranging from 1 ("not at all") to 4 ("very much").
Time to deterioration in Physical Functioning (TTDPF) in the overall population | up to approximately 37 months
  Time to deterioration in Physical Functioning (TTDPF) is defined as the time from randomization until the change from baseline reaches a clinically meaningful deterioration threshold using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Physical Functioning (QLQ-C30 PF) subscale score (EORTC IL166), where the question responses are provided on a numerical rating scale ranging from 1 ("not at all") to 4 ("very much").
Overall Pain Severity and Pain Interference as assessed by BPI-SF questionnaire in the overall population | up to approximately 37 months
  Change from baseline in Brief Pain Inventory-Short Form (BPI-SF) pain at its worse in the last 24 hours score (scale from 0 ["no pain"] to 10 ["pain as bad as you can imagine"]), pain severity (the mean of the four pain severity items each of which ranges from 0 ["no pain"] to 10 ["pain as bad as you can imagine"]) and interference domain scores (the mean of the seven pain interference items each of which ranges from 0 ["does not interfere"] to 10 ["completely interferes"]).
Plasma concentration of capivasertib derived from a population PK model in the overall population | pre dose (up to 90 minutes prior) and post dose (1 hour, 2 hours and 4 hours post dose)

OTHER OUTCOMES:
The number of participants with adverse events in the overall population | Up to approximately 46 months
  Data will include clinical observations, ECG parameters, clinical chemistry / haematology / glucose metabolism parameters and vital signs assessed as the number of participants with adverse events.
Systolic and diastolic blood pressure | Up to approximately 46 months
  millimetre of mercury (mmHg)
Pulse rate (heart rate) | Up to approximately 46 months
  Beats per minute (BPM)
Body Temperature | Up to approximately 46 months
  Celsius (°C)
Weight | Up to approximately 46 months
  Kilograms (kg)

CONTACTS AND LOCATIONS:
Locations (178):
- United States (34):
  - Research Site, Yuma, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Cerritos, California
  - Research Site, Fresno, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Aurora, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Baltimore, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Hackensack, New Jersey
  - Research Site, Albany, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Toledo, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Watertown, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Seattle, Washington
- Australia (7):
  - Research Site, Birtinya
  - Research Site, Greenslopes
  - Research Site, Kogarah
  - Research Site, North Adelaide
  - Research Site, Orange
  - Research Site, Redcliffe
  - Research Site, Wahroonga
- Belgium (3):
  - Research Site, Brasschaat
  - Research Site, Ghent
  - Research Site, Liège
- Brazil (12):
  - Research Site, Cachoeiro de Itapemirim
  - Research Site, Ijuí
  - Research Site, Itajaí
  - Research Site, Joinville
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santa Maria
  - Research Site, São José Do Rio Preto - SP
  - Research Site, São Paulo
  - Research Site, Três Lagoas
- Canada (6):
  - Research Site, Halifax, Nova Scotia
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Toronto
- Chile (2):
  - Research Site, Santiago
  - Research Site, Viña del Mar
- China (18):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jiaxing
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Yantai
  - Research Site, Zhengzhou
- Czechia (4):
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Pardubice
  - Research Site, Prague
- France (12):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Saint-Mandé
  - Research Site, Strasbourg
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Greece (5):
  - Research Site, Athens
  - Research Site, Chaïdári
  - Research Site, Marousi
  - Research Site, Pátrai
  - Research Site, Piraeus
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Szolnok
- India (4):
  - Research Site, Bikaner
  - Research Site, Meerut
  - Research Site, Mohali
  - Research Site, New Delhi
- Israel (7):
  - Research Site, Be’er Ya‘aqov
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Japan (19):
  - Research Site, Chiba
  - Research Site, Hirakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Kanazawa
  - Research Site, Kashihara-shi
  - Research Site, Kita-gun
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagoya
  - Research Site, Nakano
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Tsu
  - Research Site, Wakayama
  - Research Site, Yokohama
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Oaxaca City
  - Research Site, Zapopan
- Netherlands (2):
  - Research Site, Hoofddorp
  - Research Site, The Hague
- Poland (3):
  - Research Site, Nowa Sól
  - Research Site, Opole
  - Research Site, Wieliszew
- South Korea (4):
  - Research Site, Bukgu
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Sabadell
  - Research Site, Seville
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Edirne
  - Research Site, Izmir
  - Research Site, Şahinbey
  - Research Site, Yüreğir
- United Kingdom (8):
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, Hackensack
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home